CLINICAL TRIAL: NCT03300115
Title: Single-arm,Multi-center,Phase II Clinical Trial of the Efficacy and Safety of AC0010 in the Treatment of EGFR T790M Mutation-positive Patients With Advanded NSCLC
Brief Title: Clinical Trial of the Efficacy and Safety of AC0010 in the Treatment of EGFR T790M Patients With Advanded NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hangzhou ACEA Pharmaceutical Research Co., Ltd. (Industry)
Collaborators: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC201602AVTN03
Record Dates: First submitted 2017-09-27; First posted 2017-10-03 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Metastatic Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — abivertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AC0010 (Experimental): Each participant will be given AC0010 300mg bid.
  Interventions: Drug: AC0010

INTERVENTIONS:
Drug: AC0010 — After subjects prove eligible after screening and are enrolled, they are given AC0010 300 mg Bid (the two doses are advised to be administered at an interval of 12 hours), receive evaluation of safety indicators every 3 weeks, efficacy evaluation every 6 weeks until disease progression or intolerable toxicities or withdrawal from the trial. (If the investigator suspects disease progression, CT or MRI may be performed in advance; if the patient does not have disease progression, subsequent efficacy evaluation will proceed still according to the protocol).
  Other Names: AC0010MA

SUMMARY:
The study is a single-arm, multi-center, open-label clinical trial. The study aims to expand the sample size based on the fixed dose recommended by the results of previous dose exploration studies in order to further evaluate the study drug's efficacy and safety.

DETAILED DESCRIPTION:
The study is a single-arm, multi-center, open-label clinical trial. The study aims to expand the sample size based on the fixed dose recommended by the results of previous dose exploration studies in order to further evaluate the study drug's efficacy and safety with overall objective tumor response rate (ORR) as the primary efficacy evaluation indicator, and further evaluate subjects' duration of response (DOR), progression-free survival (PFS), disease control rate (DCR), overall survival (OS) and quality of life (QoL). Safety indicators of subjects are further evaluated through adverse events, vital signs and clinical laboratory parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years (including 18 and 75 years old).
2. Histologically or cytologically confirmed metastatic or unresectable locally advanced, recurrent non-small cell lung cancer which cannot receive radical surgery and radiotherapy.
3. The patient has at least one radio graphically (CT, MRI)measurable lesion according to the RECIST criteria for solid tumor response; long-diameter of tumor scanned by CT&MRI ≥10mm, or short-diameter of metastatic cervical lymph nodes≥15mm. With no radiotherapy and biopsy.
4. Patients without CNS metastases or asymptomatic patients with brain metastases. The number of CNS metastases focus≤2, maximum diameter <10mm.
5. Document prove EGFR mutation before treatment of EGFR TKI, or show clinical benefit after treatment of EGFR TKI (PR, CR evaluation according to RECIST or more than half-year SD duration); tumor tissue proved to be EGFR T790M positive mutation by center lab after last treatment.
6. Patients need to undergo biopsy of primary or metastatic tumor tissue and provide pathological sections to site's central lab; otherwise, the patients need to undergo biopsy of primary or metastatic tumor tissue in the screening period and provide pathological sections to the site's central laboratory.
7. Patients who have previously received first-generation EGFR-TKI (erlotinib, gefitinib, ectectin) treatment and developed resistance and are only allowed to have received one chemotherapy regimen (maintenance treatment with the same drug is allowed; but maintenance treatment with a different drug is not allowed), or are positive for primary T790M mutation but have not received treatment or have only received first-line treatment.
8. The patient must have good organ function, including meeting the laboratory test requirements at screening.
9. Patients must recover to ≤Grade 1 (CTCAE v4.03)toxicity from the previous treatment (patients with any grade of hair loss are allowed to enter the study).
10. ECOG score: 0-1 points. No deterioration in the last 2 weeks.
11. Expected survival time:> 12 weeks.
12. Patients who can cooperate with the observation of adverse events and efficacy.
13. Patients or their legal representatives have signed a written informed consent form.

Exclusion Criteria:

1. Acute hepatitis C, chronic hepatitis C and active hepatitis B (positive HBsAg; HBcAb or HBeAb positive and HBV DNA positive).
2. HIV antibody positive, or other acquired, congenital immunodeficiency disease, or a history of organ transplantation.
3. A past history of interstitial lung disease and radiation pneumonia.
4. Clinically significant abnormalities of resting ECG in rhythm, conduction and morphology, such as complete left bundle branch block, Grade II and above heart block, PR interval> 250 ms, or myocardial infarction within the past 6 months; there are risk factors leading to prolongation of QTc interval or increasing arrhythmias, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or medical history of sudden death at an age of < 40 years among the patient's first-degree relatives, and 12-lead ECG QT interval correction Fridericia method (QTcF interval)> 450 ms for male, >470ms for female.
5. The investigator judges based on safety concerns or clinical study process that the patient had any other condition that is prohibited for participation in the clinical study, such as severe infection/inflammation, intestinal obstruction, inability to swallow medication, social/psychological problems, etc.

   With clinically significant electrolyte abnormalities in laboratory tests;
6. In addition to NSCLC, patients who have been diagnosed with another and/or treatment-requiring malignant disease in recent 5 years (this exclusion criterion does not include the following circumstances: completely resected basal cell and squamous cell skin cancer, inert malignant tumor currently requiring no treatment, and any type of completely resected carcinoma in situ).

   Patients who have used high-dose glucocorticoids or other immunosuppressive agents within 1 month prior to screening.
7. Interval time between previous EGFR TKI treatment and AC0010 <8 days or 5 half-time, subject to the long time; Interval time between major surgery /radiotherapy and AC0010 <4 weeks; Patients who are using any drug known to prolong QT interval or known potent CYP3A4 enzyme inducer or inhibitor within 4 weeks before the first dose.

   Patients who have used high-dose glucocorticoids or other immunosuppressive agents within 1 month prior to screening.
8. Patients who have previously administered third-generation EGFR-TKI drugs (e.g.,AZD9291, Avitinib, CO-1686, HM61713, etc.).
9. Patients who have been registered and received the study treatment or withdrawn from the study cannot be enrolled.
10. Pregnant or lactating women.
11. Women with childbearing potential are defined as all women who are physiologically able to have a pregnancy, unless they are using an efficient contraceptive method during treatment and within 7 days after discontinuation of treatment.
12. Patients who are considered by the investigator as inappropriate to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2017-05-18 (Actual); Primary Completion 2019-06-17 (Estimated); Study Completion 2020-12-17 (Estimated)

PRIMARY OUTCOMES:
ORR(Objective Response Rate) | Every 6 weeks from time of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months.
  To assess the overall objective response rate (ORR) of AC0010 in EGFR T790M mutation-positive patients with advanced non-small cell lung cancer (NSCLC).

SECONDARY OUTCOMES:
DoR (Duration of Response) | Every 6 weeks from time of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months.
  To assess the duration of response (DOR) of AC0010 in EGFR T790M mutation-positive patients with advanced non-small cell lung cancer (NSCLC).
PFS (Progression-free survival) | Every 6 weeks from time of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months.
  To assess the progression-free survival (PFS) of AC0010 in EGFR T790M mutation-positive patients with advanced non-small cell lung cancer (NSCLC).
DCR (Disease control rate) | Every 6 weeks from time of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months.
  To assess the disease control rate (DCR) of AC0010 in EGFR T790M mutation-positive patients with advanced non-small cell lung cancer (NSCLC).
OS (Overall survival) | Every 6 weeks from time of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months.
  To assess the overall survival (OS) of AC0010 in EGFR T790M mutation-positive patients with advanced non-small cell lung cancer (NSCLC).
The lung cancer symptoms and health-related quality of life (HRQoL) | Every 3 weeks from time of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months.
  To assess the safety of AC0010 in EGFR T790M mutation-positive patients with advanced non-small cell lung cancer (NSCLC).

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wu, MD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (25):
- China (25):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Daping Hospital,Research Institute of Surgery Third Military Medical University, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Medical College of HUST, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - Shandong Cancer Hospital, Jinan, Shandong
  - Tangdu Hospital, Xi’an, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital,Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang